CLINICAL TRIAL: NCT05135026
Title: Ultrasonography and Health Education During the Antenatal Visits Among the Pregnant Women to Reduce the Unnecessary Caesarean Section in a Resource Poor Setting (Bangladesh): a Cluster Randomized Control Trial
Brief Title: Ultrasonography and Health Education Can Reduce the Unnecessary Caesarean Section in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hiroshima University (Other)
Collaborators: North South University (Other); Obstetrical and Gynaecological Society of Bangladesh (OGSB), Bangladesh (Unknown)
Responsible Party: Principal Investigator, Dr. Habiba Shirin, Principal Investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/OR-NSU/IRB/0804
Record Dates: First submitted 2021-10-29; First posted 2021-11-26 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Reduce Unnecessary Caesarean Section; Increase Institutional Delivery; Increase Antenatal Care
Keywords: Caesarean section; institutional delivery; ANC; Bangladesh

STUDY DESIGN:
Intervention Model Description: From the urban area [Dhaka Medical College & Hospital (DMCH) and Sir Salimullah Medical College & Hospital (SSMCH)], we will randomly select one hospital for intervention group and another hospital for the control group and from the rural area (Munsigonj General Hospital and Savar Upazila Health Complex), one hospital will be randomly selected as intervention site and other hospital will be selected as comparison site.
Masking Description: One research staff, who will not be involved any of the research activity of this trial, will do this randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): Usual care
- Intervention Group (IG) (Experimental): In the intervention hospitals, we will perform USG additional 2 times during the 3rd visit of 24-26 weeks and 5th visit of 34 weeks (2 USG and even more USG if needed + additional 4 ANC + Health education; pictorial flip chart showing danger sign during pregnancy and potential risks for unnecessary caesarean delivery to increase awareness for safe delivery) for all the enolled pregnant mothers.
  Interventions: Diagnostic Test: Ultrasonograpgy

INTERVENTIONS:
Diagnostic Test: Ultrasonograpgy — 2 USG in 3rd and 5th ANC visits and even more USG if needed + 4 ANC + Health education
  Other Names: Additional 4 ANC; Health Education
  Arms: Intervention Group (IG)

SUMMARY:
A caesarean section (C/S) is a surgical procedure performed to prevent difficulties during childbirth. World Health Organization considered the standard rate for the C/S would be between 10% and 15%. However, since 2000 the rate of C/S was increasing globally, and it became about twofold from 12.1% to 21.1% in 2015.

In Bangladesh, C/S continued to increase from 8% (2007) to 33% (2017). Medically unnecessary C/S was estimated about 77% of all C/S in 2018, and it was increased from 66% since 2016. In Bangladesh, unnecessary C/S observed 9.0% and 3.2% C/S done due to avoid labour pain and 5.8% for the convenience of the mother. The economic burden of each C/S is average USD 612 and unfortunately, each patient spends this amount of money from out of pocket. Aim of this study is to do ultrasonography and health education can reduce unnecessary caesarean section among pregnant women compared to control group in a resource poor setting.

Investigators will conduct this randomized controlled trial (RCT) at Dhaka and Sir Salimullah Medical College & Hospital, and two rural Upazila Health Complexes (Savar Upazila Health Complex and Munshigonj General Hospital). Investigators will randomly select one urban hospital from two urban hospitals and one rural hospital from two rural hospitals for the intervention. The other one urban and one rural hospital will be assigned as control hospitals. One research staff, who will not involve any of the research activity of this trial, will do this randomization. Pregnant mothers will be identified and recruited during their routine antenatal visits. Pregnant mothers receive 2 USG during their routine ANC visits at 1st visit of 8-12 weeks and 4th visit of 36-38 weeks. In the intervention centres, Investigators will perform additional 4 ANC visits at 20, 30, 36 and 40 weeks (total 8 visits) and USG additional 2 times during the 2nd visit of 24-26 weeks and 5th visit of 34 weeks (2 routine USG + 2 USG in 3rd and 5th ANC visits and even more USG if needed + Health education; pictorial flip chart showing danger sign during pregnancy and potential risks for unnecessary caesarean delivery to increase awareness for safe delivery) for all the enrolled pregnant mothers. In the control centres, Investigators will collect information from the pregnant mothers.

Investigators are expecting the pregnant women who will receive antenatal care with ultrasonography and health education will have reduced number of unnecessary C/S compared to control group who will not receive those.

ELIGIBILITY:
Inclusion Criteria:

1. All the pregnant mothers irrespective of age who will be attending the designated hospitals/health complex.
2. We will include all pregnant mothers who will have/have not complication to see the delivery outcome with indication of normal delivery and CS.
3. Willing to participate in the study.

Exclusion Criteria:

1. Not willing to participate.
2. Early Pregnancy with indication for C/S (co-morbidities, H/O previous C/S etc.)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant mother
Enrollment: 288 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Unnecessary C/S | 36 weeks
  Compare the reduction of the percentage of unnecessary C/S among the intervention compare to control pregnant women

SECONDARY OUTCOMES:
ANC | 36 weeks
  The rate of set-number (8 times) of ANC and post-natal (PNC) visits rates among the intervention pregnant women (how many pregnant women in IG followed the protocol.)
USG | 36 weeks
  The rate of set-number (4 times) of USG use among the intervention pregnant women (how many pregnant women in IG followed the protocol.)
Institutional (hospital and clinics) delivery compare to the home delivery | 36 weeks
  The rate of the institutional (hospital and clinics) delivery among the intervention pregnant women, compared with CG.
Delivery related complications | 36 weeks
  The reduction rate of the delivery related complications [ante partum and postpartum haemorrhage (APH, PPH)] among the intervention pregnant women, compared with CG
Rate of still birth | 36 weeks
  The reduction rate of still birth among the intervention pregnant women, compared with CG.

CONTACTS AND LOCATIONS:
Locations (1):
- DMCH, SSMC, Munshiganj General Hospital and Bogra District Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. World Health Organization 2015. WHO statement on caesarean section rates. https://apps.who.int/iris/bitstream/handle/10665/161442/WHO_RHR_15.02_eng.pdf?sequence=1 2. Boerma T, Ronsmans C, Melesse DY, Barros AJD, Barros FC, Juan L, Moller A-B, Say L, Hosseinpoor AR, Yi M, Neto DdeLR, Temmerman M. Global epidemiology of use of and disparities in caesarean sections. The Lancet, 2018; 392 (10155): 1341 DOI: 10.1016/S0140-6736(18)31928-7 3. Charvalho PdaS, Hansson BM, Stjernholm VY. Indications for increase in caesarean delivery. Reprod Health, 2019; 16, 72. https://doi.org/10.1186/s12978-019-0723-8 4. Bangladesh Demographic and Health Survey 2017-2018-key indicators.pdf [https://dhsprogram.com/pubs/pdf/PR104/PR104.pdf] 5. Save the Children International 2020. Bangladesh: 51 per cent increase in "unnecessary" C-sections in two years. [https://www.savethechildren.net/news/bangladesh-51-cent-increase-"unnecessary"-c-sections-two-years#_edn2] 6. BDHS 2014 final report[ https://dhsprogram.com/publications/publication-fr311-dhs-final-reports.cfm] 7. Infographic-unnecessary-caesarean-section.pdf[ https://www.who.int/reproductivehealth/publications/unnecessary-cs-infographics/en/] 8. Hasan F, Alam MM, Hossain MG. Associated factors and their individual contributions to caesarean delivery among married women in Bangladesh: analysis of Bangladesh demographic and health survey data. BMC Pregnancy Childbirth, 2019;19(1):433. doi:10.1186/s12884-019-2588-9 9. World Health Organization 2016. Pregnant women must be able to access the right care at the right time, says WHO. https://www.who.int/news-room/detail/07-11-2016-pregnant-women-must-be-able-to-access-the-right-care-at-the-right-time-says-who 10. Dowswell T, Carroli G, Duley L, Gates S, Gülmezoglu AM, Khan-Neelofur D, Piaggio G. Alternative versus standard packages of antenatal care for low-risk pregnancy. Cochrane Database Syst Rev. 2015;(7):CD000934 11. World Health Organization 2018. WHO recommendation on antenatal care contact schedules. https://extranet.who.int/rhl/topics/improving-health-system-performance/who-recommendation-antenatal-care-contact-schedules 12. Alland JYK, Ali H, Mehra S, LeFevre AE, Pak SE, Shaikh S, Christian P, Labrique AB. Antenatal care in rural Bangladesh: current state of costs, content and recommendations for effective service delivery. BMC Health Serv Res, 2019; 19, 861. https://doi.org/10.1186/s12913-019-4696-7 13. World Health Organization 2018. WHO recommendation on early ultrasound in pregnancy. https://extranet.who.int/rhl/topics/preconception-pregnancy-childbirth-and-postpartum-care/antenatal-care/who-recommendation-early-ultrasound-pregnancy 14. Ryan BL, Krishnan RJ, Terry A, Thind A. Do four or more antenatal care visits increase skilled birth attendant use and institutional delivery in Bangladesh? A propensity-score matched analysis. BMC Public Health, 2019;19(1):583. 15. Pervin J, Moran A, Rahman M, Razzaque A, Sibley L, Streatfield PK, Reichenbach LJ, Koblinsky M, Hruschka D, Rahman A. Association of antenatal care with facility delivery and perinatal survival - a population-based study in Bangladesh. BMC Pregnancy Childbirth, 2012;12:111. doi:10.1186/1471-2393-12-111 16. World Bank 2014. The World Bank Annual Report 2014. Washington, DC. © World Bank. https://openknowledge.worldbank.org/handle/10986/20093 License: CC BY-NC-ND 3.0 IGO. 17. Bangladesh_country_report.pdf [ https://www.who.int/pmnch/knowledge/publications/bangladesh_country_report.pdf] 18. Begum T, Ellis C, Sarker M, et al. A qualitative study to explore the attitudes of women and obstetricians towards caesarean delivery in rural Bangladesh. BMC pregnancy and childbirth, 2018;18(1):368. 19. The United Nations Children's Fund (UNICEF). Monitoring the situation of children and women. Maternal mortality, 2019. https://data.unicef.org/topic/maternal-health/maternal-mortality/ 20. Centers for Disease Control and Prevention (CDC). U.S. Department of Health & Human Services. https://www.cdc.gov/ncbddd/stillbirth/facts.html 21. Ylva Vladic Stjernholm. Caesarean section: reasons for and actions to prevent unnecessary caesareans. Open access peer-reviewed chapter. 2018. DOI: 10.5772/intechopen.76582. https://www.intechopen.com/chapters/63427 22. Charan J, Biswas T. How to calculate sample size for different study designs in medical research?. Indian J Psychol Med. 2013;35(2):121-126. doi:10.4103/0253-7176.116232
- [Derived] Shirin H, K A T M Ehsanul H, Hawlader MDH, Masud SB, Misty K, Dewan F, Moriyama M. Effectiveness of WHO-recommended antenatal care visits, ultrasonography, and health education in reducing unnecessary caesarean sections among pregnant women in Bangladesh: a hospital-based randomised controlled trial. J Glob Health. 2025 Jun 27;15:04182. doi: 10.7189/jogh.15.04182. PMID 40576427
- [Derived] Shirin H, Moriyama M, Huq KATME, Rahman MM, Masud SB, Begum RA, Misty K, Hawlader MDH. Association of Ultrasonography and Health Education during Antenatal Visits among Pregnant Women to Reduce Unnecessary Caesarean Section in Bangladesh: Study Protocol for a Cluster Randomized Control Trial. Methods Protoc. 2022 Dec 17;5(6):101. doi: 10.3390/mps5060101. PMID 36548143